CLINICAL TRIAL: NCT01838564
Title: The PediQUEST Study: Evaluation of Pediatric Quality of Life and Evaluation of Symptoms Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joanne Wolfe, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 04-321; 1K07CA096746-01 (NIH)
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Pediatric Neoplasm; Quality of Life; Outcome Assessment; Palliative Care
Keywords: Pediatric Advanced Cancer; Children; Quality of Life; Health Information technology; Patient reported outcomes
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine data collection (Active Comparator): Routine collection of patient-reported symptom and Quality of life data using PediQUEST surveys
  Interventions: Other: Routine Data collection
- Feedback of patient-reported outcomes (Experimental): Routine collection of QOL and symptom data + feedback
  Interventions: Other: Routine Data collection; Other: Feedback of patient-reported outcomes

INTERVENTIONS:
Other: Routine Data collection — Patients assigned to the control arm answered PediQUEST (PQ) surveys at most once a week and at least once a month. PQ-surveys were administered through a tablet computer if patient was at the clinic or ward or over the phone if patient was primarily at home. PQ-survey had 9 age- and respondent- adapted versions.
  Control arm participants reported their satisfaction with the PediQUEST technology twice 4th and 8th PediQUEST administration. These surveys were embedded in PediQUEST.
  Other Names: Control arm
Other: Feedback of patient-reported outcomes — Patients, parents and primary providers received printed reports summarizing patient/parent reported outcomes for last five visits. When child reported moderate-severe distress an email was automatically sent to primary providers (oncologist, nurses and psychosocial clinicians), as well as to the pain and palliative care services.
  Other Names: Feedback; Intervention arm
  Arms: Feedback of patient-reported outcomes

SUMMARY:
Over 50% of children dying from cancer still suffer from symptoms that could be effectively alleviated. The purpose of the Pediatric Quality of Life and Evaluation of Symptoms Technology (PediQUEST) Study was to evaluate whether providing feedback to families and providers about how the child is feeling improved child distress and quality of life (QoL) in children with advanced cancer.

PediQUEST is a computerized survey that asks the child and/or parents how the child has been feeling, i.e. whether the child had any physical or emotional symptoms, as well as how other aspects of life, such as school and friends, are going. After the survey is complete a report that summarizes patient/parent answers is printed. When a child reports moderate to high distress from any symptom an email is automatically sent to the primary providers (oncologist, nurse, and psycho-social clinician as well as the pain and palliative care services) alerting them about the child's distress.

In this study we evaluated whether using PediQUEST and providing printed reports to parents and providers reduced distress and improved quality of life in children with advanced cancer. In addition, we wanted to understand whether it was feasible to carry out a randomized controlled trial in children with advanced cancer. Finally, the data collected, will be used to describe the natural history of symptoms and quality of life as reported by the children.

Children enrolled in the study (or their parents) were asked to complete a PediQUEST survey at most once a week. A random half of the children received the feedback intervention, i.e. patients, parents, and providers received printed reports (and emails if the child was in distress). The other half only completed the PediQUEST surveys and did not receive reports. We analyzed data collected over 20 weeks of follow-up to see whether receiving PediQUEST reports had any effect on child distress and quality of life.

DETAILED DESCRIPTION:
Introduction: Cancer is the leading cause of nonaccidental death in childhood.(Arias et al. 2003) In spite of significant scientific progress, one quarter of children with cancer still do not survive(Greenlee et al. 2000), and over 50% experience substantial suffering that could be alleviated.(Wolfe et al. 2000a) Pediatric palliative care is now an expected standard of care and research in this field has been established as a national priority by the Institute of Medicine (IOM).(Field et al. 2003) Earlier work by our group suggested that when parents and physicians recognized at an early stage that a child had no realistic chance of cure, they were more likely to integrate elements of effective palliation into the child's care. However, this early stage concordance about prognosis was rare.(Wolfe et al. 2000b) Communication and delivery of optimal care in the advanced stages of illness is especially challenging in children.(Shelton 1999) The anticipation of losing a child and physicians' own difficulties(Saunders 1979-80; Hilden et al. 2001) may hinder discussions about poor prognosis and impact on decision-making and integration of palliative care. Thus attention to symptom management and quality of life (QoL) in children with advanced cancer may be limited.

The collection of standardized symptom and QoL data has shown to enhance physician's recognition, knowledge and accuracy in the assessment and palliation of symptoms, and to increase patient-provider discussions about QoL issues and directly improve patient's QoL.(Detmar et al. 2002; Taenzer et al. 2000; Velikova et al. 2004) Whether these findings are applicable to children remains to be established.

One of the obstacles to routine symptom and QoL assessment in children is the need of developmentally adapted(Eiser et al. 2001b; Eiser et al. 2001c; Hain 1997) and parent-proxy tools(Eiser et al. 2001a), making the paper and pencil format extremely impractical. Computerized surveys offered a potential solution. Patient acceptance of such devices has been found to be high.(Buxton et al. 1998; Velikova et al. 2002; Velikova et al. 1999; Velikova et al. 2001) Our current project -the PediQUEST Study- consists of a pilot for a randomized controlled trial (RCT) aimed at assessing the effect of routinely reporting symptom and QoL data. We will use an innovative data collection strategy: a hand-held computer devise, the Pediatric Quality of Life and Evaluation of Symptoms Technology (PediQUEST) that readily administers a user-appropriate survey instrument and generates reports summarizing how the patient feels.

As far as we are aware of, this will be the first RCT conducted in children with advanced cancer to evaluate a palliative care intervention. Given the challenges with doing research in this population, we propose to simultaneously focus on several goals.

Aims: Aim 1: (Feasibility study) Assess the feasibility of conducting a randomized controlled supportive care trial (RCT) in children with advanced cancer. Aim 2: (PediQUEST Evaluation) Preliminarily assess the effect of routinely feeding back QoL and symptom data to families and primary oncologists, and alerting supportive care teams about highly distressing symptoms. Aim 3: (Descriptive study) Prospectively explore determinants of child's suffering and parental-physician discordance regarding prognosis and treatment goals in children with advanced cancer.

Design: Aim 1: Cohort survey study; Aim 2: Pilot prospective RCT; Aim 3: Cohort study embedded in an RCT.

Setting: Three large US pediatric cancer centers. Subjects: 104 children 2-years old and above with advanced cancer and their parents were enrolled between December 2004 and June 2009.

Follow-up: Patients were initially followed up for 9 months or until death whatever occurred first. However, an interim analysis of the first 29 patients showed that 75% were alive at nine months, suggesting the enrollment of a healthier cohort. We therefore changed the follow-up period to 3 months with the option of multiple re-enrollments until the end of data collection (December 2009) or death.

Methods:

Feasibility study: All subjects approached for enrollment were invited to complete a one-time paper and pencil "Consent survey" regardless of their decision about whether to participate. All enrolled subjects were asked to complete a paper and pencil "Participation survey" after completing the study or dropping-out in order to explore determinants of attrition.

PediQUEST Evaluation and Descriptive studies: Symptom and QOL scores were tracked up to once a week. Surveys were embedded in the PediQUEST system and administered through tablet computers.

Participants' recruitment: Eligible children were identified through daily review of clinic roster with clinic staff including nurses, oncologists and/or nurse practitioners and verified with the patient's primary oncologist using a checklist sent over email. If after being introduced to the study and having had the opportunity to ask questions, child and parent(s) were willing to participate, parent(s) were asked to review and sign the informed permission/assent document covering the parent(s) and child's participation. A provider's completion of the eligibility checklist will indicate informed consent of providers.

Study Instruments:

1. PediQUEST survey (PQ-Survey): assessed symptoms, quality of life, and overall sickness. Nine survey versions were developed to allow for consistent measurement across the age ranges and respondents. Self-report started at 5 years of age; children aged 5 to 12 years answered shorter, age-adapted questionnaires which were complemented with additional parental questionnaires; teens answered a full self-report questionnaire. Parents of children between 2 and 4 years old answered a full survey on their child's behalf. If a child did not feel well, parents could complete the full questionnaire on their behalf. PQ-Surveys were pilot tested in 15 patients showing good acceptability and comprehensibility. PQ-surveys used four tools: 1) PQ-Memorial Symptom Assessment Scale (MSAS), adapted from previously validated child(Collins et al. 2000; Collins et al. 2002) and proxy(Drake et al. 2003) MSAS, measures frequency, severity and distress for 24 symptoms; 2) Pediatric Quality of Life Inventory (PedsQL), a 22-item health related quality of life instrument;(Seid et al. 1999; Varni et al. 2002; Varni et al. 2003) 3) Faces Pain Scale Revised (a faces pain scale, used to measure current pain intensity);(Hicks et al. 2001) 4) Sickness VAS scale (overall sickness measure created ad hoc).
2. Survey about Caring for Children with Cancer (SCCC): In addition, parent and physician perspectives regarding prognosis and treatment goals were collected at baseline and then every 3 months using a paper-and-pencil survey SCCC, adapted from our survey for bereaved parents.(Wolfe et al. 2000b)
3. Post death survey: If patients died within the study period parents were invited to complete a post-death survey at least four months following the death to assess distress during the last month of life and retrospective perspectives regarding the overall quality of care.
4. Satisfaction Surveys: Child and parent surveys were adapted from existing questionnaires.(Grogan et al. 1995; McCusker 1984; Weaver et al. 1993) Satisfaction with PQ technology was assessed using seven items for children eight years old and above and 11 items for parents. Surveys were embedded in the PediQUEST system and administered at fourth and eighth PediQUEST administration. A survey evaluating participant's satisfaction with the PediQUEST intervention (see below) was administered concurrently (eight items (parents), five items (children eight years old and above)) to all intervention participants. Provider satisfaction with the PQ intervention, and perceived usefulness of the PQ-system was assessed through an online survey administered at the end of data collection.

Intervention: Patients were randomly allocated to receive routine feedback about symptoms and QOL. The feedback intervention had two components: (i) PQ-reports: printed reports were made available to providers (inserted in charts before the visit) and families (handed immediately after survey completion at clinic or ward). PQ-reports consisted of bar plots of PedsQL and MSAS symptom scores from current and four prior administrations, a summary highlighting changes since last report, and a list of available resources for symptom control (for families), or generic pain management recommendations (for providers). Training on how to interpret PQ-reports was offered to families at enrollment and on an annual basis to providers; (ii) PQ emails: were automatically generated if PQ-MSAS individual symptom scores were ≥70, or if on two consecutive administrations the patient or parent reported a score of ≥70 for any frequency, severity or distress item, or a PedsQL total score ≤ 40. E-mails were sent to primary providers (oncologist, nurse, and psychosocial clinician), the local palliative care service, and, when pain was reported, the pain service (or equivalent). No instructions were imparted on how to respond to emails. Families and providers of patients in the control arm of the study did not receive feedback reports. The allocation process was embedded in PediQUEST and blinded to investigators until the patient completed the first survey. Because of the nature of the intervention this was an open label study. As a token of our appreciation, small non-monetary incentives were provided to children, parents, and providers.

Outcomes: This study explores the feasibility of conducting an RCT assessing a supportive care intervention in children with advanced cancer (aim 1). It also provides estimates of consent and attrition rates, its determinants, and the burden associated with repeated measurements. In addition, this pilot study will preliminarily assess the impact of feedback on child's distress and quality of life. Main outcomes of this efficacy study (aim 2) are presented below. This pilot study will render sufficient data for accurate sample size calculation for future studies and serve to explore determinants of suffering in children with advanced cancer (aim 3).

Statistical Analysis:

PediQUEST Evaluation (Aim 2): To assess the effect of PediQUEST, the proportion of patients with unrelieved symptoms in each arm will be compared using odds ratios and associated chi-square tests. To assess the progression of reported levels of child's distress and QOL trends, we will run a mixed effects model that assumes a linear trend in the outcome over 20 weeks of follow up for each subject. The model will examine the difference in the average trend over time (slope) between the intervention and control group by including a fixed effect term that represents the interaction of treatment status and time since study entry. Lack of difference between slope coefficients will support the null hypothesis of no effect by the intervention. Single point secondary outcomes will be analyzed by comparing both arms with a t test or Wilcoxon rank-sum test for continuous outcomes and odds ratios and associated chi-square tests for proportions.

Sample Size and Power Calculations A formal sample size estimation was not possible given the lack of data on distribution of scores in an advanced cancer population or their variation over time. For this reason we originally proposed to recruit 120 patients and their parents, a sample size driven by practical rather than statistical considerations that would serve as a basis for future sample size calculations. We estimated that 60 subjects per arm would allow for an adequate balance between arms and likely provide sufficient power to detect large clinical effects for single point measurements.

ELIGIBILITY:
Inclusion Criteria:

* Children >=2-years old with at least a 2-week history of progressive, recurrent, or non-responsive cancer of any type or decision not to pursue cancer directed therapy.
* Child's parent must have spoken and written command of English or Spanish.
* Child's parent must have the ability to understand and complete self-administered surveys.

Exclusion Criteria:

* Patients who have an isolated relapsed solid tumor treated with surgery or radiation alone.
* Patients with hematological malignancies who have achieved remission after the first induction attempt, whose treatment plan includes their first Stem Cell Transplant (SCT), and have an identified donor (must meet all 3 criteria to be excluded).
* Patients who are not regular patients at one of the two participating institutions.
* Foster parents who do not have legal guardianship.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2004-11; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Child Distress - unrelieved symptoms | 20 weeks
  Child distress-unrelieved symptoms will be assessed through the proportion of patients with unrelieved symptoms (any symptom/s reported as causing moderate to high distress or FPS-R score >=8 in 2 consecutive PediQUEST evaluations)
Trends of PedsQL Total Scores | 20 weeks
  Trends of PedsQL total scores over time. PedsQL is a continuous variable (Range: 0-100. 100 highest quality of life).
Trends of MSAS total scores | 20 weeks
  Trends of MSAS total score over time(MSAS total score is a continuous variable; range: 0-100. 100 worst).
Trends of MSAS physical scores | 20 weeks
  Trends over time of MSAS physical subscale scores (MSAS physical subscale score is a continuous variable. Range: 0-100. 100 highly symptomatic.)
Trends of MSAS psychological scores | 20 weeks
  Trends over time of MSAS psychological subscale scores (MSAS psychological subscale scores is a continuous variable. Range: 0-100. 100 highly symptomatic.)
Trends of PedsQL Physical Subscale Scores | 20 weeks
  Trends of PedsQL physical subscale scores over time. PedsQL physical score is a continuous variable (Range: 0-100. 100 highest quality of life).
Trends of PedsQL Emotional Subscale Scores | 20 weeks
  Trends of PedsQL emotional subscale scores over time. PedsQL emotional score is a continuous variable (Range: 0-100. 100 highest quality of life).

SECONDARY OUTCOMES:
Parental distress over time | 20 weeks
  Trends in Kessler-6 scores (general psychological distress scale) over 20 weeks. Continuous variable. Range:0-24 (24 is high distress).
Patterns of care - Referrals to support services | 20 weeks
  N° of referrals to support services (Psychiatry service, Pastoral Care): continuous variable.
Patterns of care - Chemotherapy during last month of life | 20 weeks
  Proportion of patients receiving chemotherapy during the last month of life
Patterns of care - Use of hospice/home care | 20 weeks
  Proportion of patients receiving home care assistance or hospice care
Patterns of care - Time of documentation of prognosis discussions | 20 weeks
  Time of documentation (N° of days before death) of discussions about prognosis
Patterns of care - Time of documentation of resuscitation status | 20 weeks
  Time of documentation (N° of days before death) of discussions about resuscitation status
Patterns of care - Ventilatory assistance in last day of life | 20 weeks
  Proportion of patients who were intubated in the last 24 hrs of life.
Patterns of care - Hospital deaths | 20 weeks
  Proportion of patients who died at the hospital

OTHER OUTCOMES:
Satisfaction with PediQUEST | At 4th PediQUEST administration
  Satisfaction with the technology and with the feedback system will be assessed twice at the fourth and eight PediQUEST administration. Specifically we will assess consumers'impressions about the technology, easiness of use, relevance.
  Among those receiving the feedback intervention we also assessed whether reports helped parents understand their children's feelings better, facilitated communication with doctors and overall satisfaction with the technology and feedback.
  Finally, we also assessed providers satisfaction with feedback reports including their impression about the reports and whether reports affected their behaviors regarding symptom management.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Wolfe, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Philapdelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Arias E, MacDorman MF, Strobino DM, Guyer B. Annual summary of vital statistics--2002. Pediatrics. 2003 Dec;112(6 Pt 1):1215-30. doi: 10.1542/peds.112.6.1215. PMID 14654589
- [Background] Buxton J, White M, Osoba D. Patients' experiences using a computerized program with a touch-sensitive video monitor for the assessment of health-related quality of life. Qual Life Res. 1998 Aug;7(6):513-9. doi: 10.1023/a:1008826408328. PMID 9737141
- [Background] Collins JJ, Byrnes ME, Dunkel IJ, Lapin J, Nadel T, Thaler HT, Polyak T, Rapkin B, Portenoy RK. The measurement of symptoms in children with cancer. J Pain Symptom Manage. 2000 May;19(5):363-77. doi: 10.1016/s0885-3924(00)00127-5. PMID 10869877
- [Background] Collins JJ, Devine TD, Dick GS, Johnson EA, Kilham HA, Pinkerton CR, Stevens MM, Thaler HT, Portenoy RK. The measurement of symptoms in young children with cancer: the validation of the Memorial Symptom Assessment Scale in children aged 7-12. J Pain Symptom Manage. 2002 Jan;23(1):10-6. doi: 10.1016/s0885-3924(01)00375-x. PMID 11779663
- [Background] Detmar SB, Muller MJ, Schornagel JH, Wever LD, Aaronson NK. Health-related quality-of-life assessments and patient-physician communication: a randomized controlled trial. JAMA. 2002 Dec 18;288(23):3027-34. doi: 10.1001/jama.288.23.3027. PMID 12479768
- [Background] Drake R, Frost J, Collins JJ. The symptoms of dying children. J Pain Symptom Manage. 2003 Jul;26(1):594-603. doi: 10.1016/s0885-3924(03)00202-1. PMID 12850642
- [Background] Eiser C, Morse R. Can parents rate their child's health-related quality of life? Results of a systematic review. Qual Life Res. 2001;10(4):347-57. doi: 10.1023/a:1012253723272. PMID 11763247
- [Background] Eiser C, Morse R. Quality-of-life measures in chronic diseases of childhood. Health Technol Assess. 2001;5(4):1-157. doi: 10.3310/hta5040. PMID 11262421
- [Background] Eiser C, Morse R. A review of measures of quality of life for children with chronic illness. Arch Dis Child. 2001 Mar;84(3):205-11. doi: 10.1136/adc.84.3.205. PMID 11207164
- [Background] Institute of Medicine (US) Committee on Palliative and End-of-Life Care for Children and Their Families; Field MJ, Behrman RE, editors. When Children Die: Improving Palliative and End-of-Life Care for Children and Their Families. Washington (DC): National Academies Press (US); 2003. Available from http://www.ncbi.nlm.nih.gov/books/NBK220818/ PMID 25057608
- [Background] Greenlee RT, Murray T, Bolden S, Wingo PA. Cancer statistics, 2000. CA Cancer J Clin. 2000 Jan-Feb;50(1):7-33. doi: 10.3322/canjclin.50.1.7. PMID 10735013
- [Background] Grogan S, Conner M, Willits D, Norman P. Development of a questionnaire to measure patients' satisfaction with general practitioners' services. Br J Gen Pract. 1995 Oct;45(399):525-9. PMID 7492421
- [Background] Hain RD. Pain scales in children: a review. Palliat Med. 1997 Sep;11(5):341-50. doi: 10.1177/026921639701100503. PMID 9472590
- [Background] Hilden JM, Emanuel EJ, Fairclough DL, Link MP, Foley KM, Clarridge BC, Schnipper LE, Mayer RJ. Attitudes and practices among pediatric oncologists regarding end-of-life care: results of the 1998 American Society of Clinical Oncology survey. J Clin Oncol. 2001 Jan 1;19(1):205-12. doi: 10.1200/JCO.2001.19.1.205. PMID 11134214
- [Background] McCusker J. Development of scales to measure satisfaction and preferences regarding long-term and terminal care. Med Care. 1984 May;22(5):476-93. doi: 10.1097/00005650-198405000-00011. PMID 6425580
- [Background] Saunders CM. A comparison of adult bereavement in the death of a spouse, child, and parent. Omega 1979-80; 10:302-22
- [Background] Seid M, Varni JW, Rode CA, Katz ER. The Pediatric Cancer Quality of Life Inventory: a modular approach to measuring health-related quality of life in children with cancer. Int J Cancer Suppl. 1999;12:71-6. doi: 10.1002/(sici)1097-0215(1999)83:12+3.0.co;2-5. PMID 10679874
- [Background] Shelton TL. Family-centered care in pediatric practice: when and how? J Dev Behav Pediatr. 1999 Apr;20(2):117-9. doi: 10.1097/00004703-199904000-00008. No abstract available. PMID 10219691
- [Background] Taenzer P, Bultz BD, Carlson LE, Speca M, DeGagne T, Olson K, Doll R, Rosberger Z. Impact of computerized quality of life screening on physician behaviour and patient satisfaction in lung cancer outpatients. Psychooncology. 2000 May-Jun;9(3):203-13. doi: 10.1002/1099-1611(200005/06)9:33.0.co;2-y. PMID 10871716
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Background] Varni JW, Burwinkle TM, Seid M, Skarr D. The PedsQL 4.0 as a pediatric population health measure: feasibility, reliability, and validity. Ambul Pediatr. 2003 Nov-Dec;3(6):329-41. doi: 10.1367/1539-4409(2003)0032.0.co;2. PMID 14616041
- [Background] Velikova G, Booth L, Smith AB, Brown PM, Lynch P, Brown JM, Selby PJ. Measuring quality of life in routine oncology practice improves communication and patient well-being: a randomized controlled trial. J Clin Oncol. 2004 Feb 15;22(4):714-24. doi: 10.1200/JCO.2004.06.078. PMID 14966096
- [Background] Velikova G, Brown JM, Smith AB, Selby PJ. Computer-based quality of life questionnaires may contribute to doctor-patient interactions in oncology. Br J Cancer. 2002 Jan 7;86(1):51-9. doi: 10.1038/sj.bjc.6600001. PMID 11857011
- [Background] Velikova G, Wright EP, Smith AB, Cull A, Gould A, Forman D, Perren T, Stead M, Brown J, Selby PJ. Automated collection of quality-of-life data: a comparison of paper and computer touch-screen questionnaires. J Clin Oncol. 1999 Mar;17(3):998-1007. doi: 10.1200/JCO.1999.17.3.998. PMID 10071295
- [Background] Velikova G, Wright P, Smith AB, Stark D, Perren T, Brown J, Selby P. Self-reported quality of life of individual cancer patients: concordance of results with disease course and medical records. J Clin Oncol. 2001 Apr 1;19(7):2064-73. doi: 10.1200/JCO.2001.19.7.2064. PMID 11283140
- [Background] Weaver MJ, Ow CL, Walker DJ, Degenhardt EF. A questionnaire for patients' evaluations of their physicians' humanistic behaviors. J Gen Intern Med. 1993 Mar;8(3):135-9. doi: 10.1007/BF02599758. PMID 8455109
- [Background] Wolfe J, Grier HE, Klar N, Levin SB, Ellenbogen JM, Salem-Schatz S, Emanuel EJ, Weeks JC. Symptoms and suffering at the end of life in children with cancer. N Engl J Med. 2000 Feb 3;342(5):326-33. doi: 10.1056/NEJM200002033420506. PMID 10655532
- [Background] Wolfe J, Klar N, Grier HE, Duncan J, Salem-Schatz S, Emanuel EJ, Weeks JC. Understanding of prognosis among parents of children who died of cancer: impact on treatment goals and integration of palliative care. JAMA. 2000 Nov 15;284(19):2469-75. doi: 10.1001/jama.284.19.2469. PMID 11074776
- [Derived] Rosenberg AR, Orellana L, Ullrich C, Kang T, Geyer JR, Feudtner C, Dussel V, Wolfe J. Quality of Life in Children With Advanced Cancer: A Report From the PediQUEST Study. J Pain Symptom Manage. 2016 Aug;52(2):243-53. doi: 10.1016/j.jpainsymman.2016.04.002. Epub 2016 May 21. PMID 27220948
- [Derived] Wolfe J, Orellana L, Ullrich C, Cook EF, Kang TI, Rosenberg A, Geyer R, Feudtner C, Dussel V. Symptoms and Distress in Children With Advanced Cancer: Prospective Patient-Reported Outcomes From the PediQUEST Study. J Clin Oncol. 2015 Jun 10;33(17):1928-35. doi: 10.1200/JCO.2014.59.1222. Epub 2015 Apr 27. PMID 25918277
- [Derived] Dussel V, Orellana L, Soto N, Chen K, Ullrich C, Kang TI, Geyer JR, Feudtner C, Wolfe J. Feasibility of Conducting a Palliative Care Randomized Controlled Trial in Children With Advanced Cancer: Assessment of the PediQUEST Study. J Pain Symptom Manage. 2015 Jun;49(6):1059-69. doi: 10.1016/j.jpainsymman.2014.12.010. Epub 2015 Jan 30. PMID 25640275
- [Derived] Wolfe J, Orellana L, Cook EF, Ullrich C, Kang T, Geyer JR, Feudtner C, Weeks JC, Dussel V. Improving the care of children with advanced cancer by using an electronic patient-reported feedback intervention: results from the PediQUEST randomized controlled trial. J Clin Oncol. 2014 Apr 10;32(11):1119-26. doi: 10.1200/JCO.2013.51.5981. Epub 2014 Mar 10. PMID 24616307